CLINICAL TRIAL: NCT01290302
Title: Blinded Cross-over Bioequivalence Trial of Luitpold Azacitidine Versus Vidaza® in Patients With Myelodysplastic Syndrome, Myelofibrosis, Chronic Myeloid Leukemia or Chronic Lymphocytic Leukemia
Brief Title: Blinded Cross-Over Bioequivalence (BE) Trial of Luitpold Azacitidine vs Vidaza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1AZA10001
Record Dates: First submitted 2011-01-10; First posted 2011-02-07 (Estimated); Results first posted 2025-05-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-11

CONDITIONS: Myelodysplastic Syndrome; Myelofibrosis; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Azacitidine; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Luitpold Azacitidine first, then Vidaza® (Experimental): Participants first received Luitpold Azacitidine subcutaneously (SC) on Day 1. After a washout period of 24 hours, they then received Vidaza on Day 2.
  Interventions: Drug: Luitpold Azacitidine
- Vidaza® first, then Luitpold Azacitidine (Active Comparator): Participants first received Vidaza subcutaneously (SC) on Day 1. After a washout period of 24 hours, they then received Luitpold Azacitidine on Day 2.
  Interventions: Drug: Vidaza®

INTERVENTIONS:
Drug: Luitpold Azacitidine — Subcutaneous (SC) at a dose of 75 mg/m^2 per day on days 1 and 2 of a treatment cycle
  Other Names: Single use vials containing 100 mg azacitidine/vials,.The formulation contained mannitol as an excipient. Lot 090035 and Lot 120011
  Arms: Luitpold Azacitidine first, then Vidaza®
Drug: Vidaza® — Subcutaneous (SC) at a dose of 75 mg/m^2 per day on days 1 and 2 of a treatment cycle
  Other Names: Vidaza (azacitidine for injection), Celegene Corporation, commercially available formulation. The formulation contained mannitol as a excipient. Lot 91096A
  Arms: Vidaza® first, then Luitpold Azacitidine

SUMMARY:
The purpose of this study is to assess the bioequivalence of subcutaneous Vidaza® and subcutaneous Luitpold Azacitidine pharmacokinetics and to assess the comparative safety of subcutaneous Vidaza® versus subcutaneous Luitpold Azacitidine.

DETAILED DESCRIPTION:
To assess the bioequivalence of Vidaza® and Luitpold Azacitidine pharmacokinetics, in terms of Maximal Concentration (Cmax), Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC 0-t), and Area Under the Curve From Time Zero Extrapolated to Infinity (AUC 0-∞), following SC administration.

To assess the comparative safety of Vidaza® versus Luitpold Azacitidine during the 2 day study period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures.
* Patients with one of the following - myelodysplastic syndrome of the following French-American- British (FAB) subtypes: refractory anemia (RA), RA with ringed sideroblasts (if accompanied by neutropenia, or thrombocytopenia, or requiring transfusion), RA with excess of blasts (RAEB), RAEB in transformation (RAEB-T), or chronic myelomonocytic leukemia (CMMoL); myelofibrosis; chronic myeloid leukemia; or chronic lymphocytic leukemia who's physician feels should receive azacitidine.
* Male or female patients aged at least 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Life expectancy > or = to 3 months.
* Adequate organ function, including the following: Hepatic - Total bilirubin < or = to 1.5 x the upper limit of normal (ULN), aspartate transaminases (AST) and alanine transaminases (ALT) < or = to 2 x ULN and Renal - Serum creatinine < or = to 1.5 x ULN.
* Female patients of child-bearing potential must have a negative pregnancy test and must be using at least one form of contraception as approved by the Investigator for 4 weeks prior to the study and 4 months after the last dose of azacitidine.
* Male patients must use a form of barrier contraception approved by the investigator during the study and for 4 months after the last dose of azacitidine.

Exclusion Criteria:

* Hypersensitivity to azacitidine or mannitol.
* Anticipated need for red blood cells (RBC) or platelet transfusion 2 days prior to or up to 2 days after treatment initiation.
* Chemotherapy (excluding previous azacitidine treatment) or radiotherapy within 4 weeks of randomization (6 weeks for nitrosoureas or mitomycin C).
* Significant electrophysical abnormalities in pre-trial EKG.
* Present history of locally advanced or metastatic malignant disease or leukemia.
* Use of recreational drugs or history of drug addiction, within the prior 6 months.
* Known history of a positive hepatitis screen, including hepatitis B surface antigens or hepatitis C virus (HCV) antibodies.
* Known history of HIV or syphilis.
* History of clinically significant adverse events due to chemotherapy, radiotherapy or investigational agents.
* Presence of an advanced malignant hepatic tumor.
* Presence of an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders.
* Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patients compliance.
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry.
* Pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Perno, MD,PhD, Study Director — Medical Director
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-eight subjects were randomized, 33 subjects were treated, and 33 subjects were analyzed for safety and pharmacokinetics (PK)
Period: Overall Study
Arm/Group | Luitpold Azacitidine First, Then Vidaza® | Vidaza® First, Then Luitpold Azacitidine
Started | 19 | 19
Treated and Analyzed | 15 | 18
Completed | 15 | 17
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Expiration of time for screening window | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luitpold Azacitidine First, Then Vidaza® | Vidaza® First, Then Luitpold Azacitidine | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (14.66) | 68.4 (10.79) | 65.7 (12.84)
Age, Customized [Median (Full Range); unit: Years] | 65 [24 to 85] | 68.5 [45 to 85] | 67 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 33
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
  Poland | 10 | 12 | 22
Height [Mean (Standard Deviation); unit: cm] | 167.12 (9.117) | 167.51 (9.797) | 167.34 (9.348)
Height [Median (Full Range); unit: cm] | 168 [153 to 190.5] | 165.85 [149.9 to 185] | 167 [149.9 to 190.5]
Weight [Mean (Standard Deviation); unit: kg] | 76.18 (19.277) | 73.92 (10.553) | 74.95 (14.935)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.04 (4.895) | 26.48 (4.182) | 26.73 (4.456)
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.61 [20 to 35.2] | 25.73 [17.8 to 34.9] | 26.22 [17.8 to 35.2]
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.86 (0.248) | 1.85 (0.158) | 1.85 (0.201)
Body Surface Area [Median (Full Range); unit: m^2] | 1.85 [1.5 to 2.5] | 1.89 [1.5 to 2.1] | 1.86 [1.5 to 2.5]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) From Time Zero to the Time of Last Quantifiable Concentration (AUC 0-t)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; AUC 0-t is defined as AUC from time 0 to the last data point
Time Frame: 0.125, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, and 10 hours after dosing on days 1 and 2.
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Luitpold Azacitidine: Luitpold Azacitidine given on Day 1 or Day 2.
- Vidaza®: Vidaza given on Day 1 or Day 2
Arm/Group | Luitpold Azacitidine | Vidaza®
Number analyzed (Participants) | 33 | 33
ng*hr/mL | 1065 (29.3) | 1024 (43.6)

2. Primary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinity (AUC 0-∞)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC 0-∞ is defined as area under the concentration vs. time curve from zero to infinity.
Time Frame: 0.125, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, and 10 hours after dosing on days 1 and 2
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Luitpold Azacitidine | Vidaza®
Number analyzed (Participants) | 33 | 33
ng*hr/mL | 1097 (28.8) | 1041 (43.1)

3. Primary Outcome: Observed Maximal Concentration (Cmax)
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: 0.125, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, and 10 hours after dosing on days 1 and 2
Population: Intent to treat
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Luitpold Azacitidine | Vidaza®
Number analyzed (Participants) | 33 | 33
ng/mL | 749 (35.9) | 854 (77.1)

ADVERSE EVENTS:
Time Frame: 2 days
Description: An adverse event was defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Luitpold Azacitidine | Vidaza®
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 10/33 | 12/33
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luitpold Azacitidine (N=33) | Vidaza® (N=33)
Fatigue (General disorders) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Injection site hematoma (General disorders) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Blood and lymphatic system disorders (Investigations) | 0 (0) | 2 (2)
Anemia (Investigations) | 1 (1) | 1 (1)
Neutropenia (Investigations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pseudohyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes